CLINICAL TRIAL: NCT00125164
Title: Recombinant Human Insulin-Like Growth Factor (rhIGF-1) Treatment of Prepubertal Children With Growth Failure Associated With Primary IGF-1 Deficiency: A Phase 3, Randomized, Open Label, Observation-Controlled, Multicenter, Parallel-Dose Comparison Trial
Brief Title: Prepubertal Children With Growth Failure Associated With Primary Insulin-Like Growth Factor-1 (IGF-1) Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS301; 2019-001020-36 (EudraCT Number)
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Growth Disorders; Insulin-Like Growth Factor-1 Deficiency
Keywords: Primary IGF-1 Deficiency
MeSH Terms: conditions — Growth Disorders | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Untreated (No Intervention): Observational Group
- 40 μg/kg BID (twice daily dosing) (Experimental): Injection of rhIGF-1 40 μg/kg BID. Per protocol amendment these subjects were reassigned to receive 120 μg/kg BID. Due to the dose change, the efficacy results for these subjects were analysed in a separate subanalysis. For all outcome measures, mean and standard deviations were not calculated for this arm.
  Interventions: Drug: rhIGF-1 (mecasermin, Tercica, Inc.)
- 80 μg/kg BID (twice daily dosing) (Experimental): Injection of rhIGF-1 80 μg/kg BID
  Interventions: Drug: rhIGF-1 (mecasermin, Tercica, Inc.)
- 120 μg/kg BID (twice daily dosing) (Experimental): Injection of rhIGF-1 120 μg/kg BID
  Interventions: Drug: rhIGF-1 (mecasermin, Tercica, Inc.)

INTERVENTIONS:
Drug: rhIGF-1 (mecasermin, Tercica, Inc.) — Twice Daily Injection
  Arms: 120 μg/kg BID (twice daily dosing); 40 μg/kg BID (twice daily dosing); 80 μg/kg BID (twice daily dosing)

SUMMARY:
This study is intended to determine whether twice daily weight based dosing with recombinant human insulin-like growth factor (rhIGF-1) will safely and effectively increase the growth of prepubertal children with short stature associated with low IGF-1 levels but who produce sufficient growth hormone (GH). Subjects will be randomized to either an observation arm or to active treatment.

DETAILED DESCRIPTION:
Prepubertal growth failure associated with primary IGF-1 deficiency (IGFD). Primary IGFD is a term that has been used to describe patients with intrinsic cellular defects in GH action. In this protocol, primary IGFD is defined as short stature (height standard deviation score[SDS]<-2 below the mean for age and gender), low serum IGF-1 (IGF-1 SDS <-2 below the mean for age and gender), and levels of growth hormone (GH) that are normal (≥7ng/mL) after a GH stimulation test. Primary IGFD is believed to result from a lower than normal ability to produce IGF-1 when exposed to normal levels of GH, i.e., a type of GH insensitivity or GH resistance.

This trial is one year, randomized, open label, observation-controlled, parallel-dose comparison efficacy and safety study conducted in approximately 40 centers across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age ≥ 3 and chronological or bone age less than or equal to 11 years inclusive in girls;
* Chronological age ≥ 3 and chronological or bone age less than or equal to 12 years inclusive for boys
* Prepubertal
* Height SD score of < -2
* IGF-1 SD score of < -2

Exclusion Criteria:

* Prior treatment with rhGH, rhIGF-1, or other growth-influencing medications
* Growth failure associated with other identifiable causes (e.g., syndromes, chromosomal abnormality)
* Chronic illness such as diabetes, cystic fibrosis, etc.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen (formerly Tercica), Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 14 March 2004. Study completion Date: 02 July 2008. 44 investigators screened subjects; 14 did not enroll any subjects. 137 subjects were enrolled. Consent for one randomized subject was withdrawn prior to any study measurements. This subject was excluded from all analyses.
Pre-assignment Details: Subject screening consisted of three staged clinic visits over 6 weeks, including a medical history, complete physical examination, IGF-1 measurements, a Growth Hormone (GH) stimulation test, and an IGF-1 generation test.
Period: Overall Study
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Started | 25 | 16 | 44 | 51
Completed | 23 | 16 | 40 | 45
Not Completed | 2 | 0 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing) | Total
Number analyzed (Participants) | 25 | 16 | 44 | 51 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (2.4) | 7.6 (2.4) | 7.7 (2.4) | 7.6 (2.7) | 7.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14 | 8 | 36
  Male | 15 | 12 | 30 | 43 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1 | 2 | 4
  Black | 0 | 0 | 0 | 2 | 2
  Hispanic | 2 | 0 | 4 | 4 | 10
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 1 | 1
  White | 22 | 16 | 38 | 41 | 117
  Other | 0 | 0 | 1 | 1 | 2
Stratum [Number; unit: participants] — Please note that SD is a standard term used in growth studies and represents Standard Deviations calculated as the patient value minus the mean divided by the standard deviation. Standard Deviation Scores vary depending on the age and sex of the child.
  participants
    Height Standard Deviation Score < -2.6 | 13 | 8 | 25 | 30 | 76
    Height Standard Deviation Score >= -2.6 | 12 | 8 | 19 | 21 | 60
Height Standard Deviation (SD) Score [Mean (Standard Deviation); unit: SD] — Please note that SD is a standard term used in growth studies and represents Standard Deviations calculated as the patient value minus the mean divided by the standard deviation. Standard Deviation Scores vary depending on the age and sex of the child.
  SD | -2.8 (0.7) | -2.6 (0.6) | -2.7 (0.5) | -2.9 (0.8) | -2.8 (0.7)
IGF-1 Standard Deviation (SD) Score [Mean (Standard Deviation); unit: SD] — Please note that Standard Deviation (SD) Score is a term used in growth studies. The SD Score is calculated as the patient value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child.
  SD | -2.6 (0.7) | -2.8 (0.8) | -2.6 (0.7) | -3.0 (0.8) | -2.8 (0.8)
Maximum Stimulated Growth Hormone [Mean (Standard Deviation); unit: ng/mL] — Growth Hormone Stimulation Test results expressed in ng/mL
  ng/mL | 17.0 (6.5) | 16.9 (6.2) | 17.8 (9.0) | 20.7 (16.8) | 18.6 (12.1)
Weight [Mean (Standard Deviation); unit: Kg] | 17.8 (4.6) | 18.5 (4.7) | 19.4 (5.4) | 18.5 (5.7) | 18.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity During the First Year - Intent to Treat (ITT)Population
Description: Height to be measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. Reposition subject between each measurement.
Time Frame: Measured at baseline and at one year
Population: A modified intention-to-treat population consisting of all randomized subjects in the untreated control, 80 and 120 µg/kg BID groups with a baseline height measurement and at least one on-treatment height measurement. Subjects assigned to 40 μg/kg BID arm were excluded from the analysis due to the dose change to 120 μg/kg BID.
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 22 | 0 | 42 | 49
cm/yr | 5.2 (1.0) |  | 6.9 (1.0) | 7.7 (1.5)
Statistical Analysis 1: Comparison: Untreated vs 80 μg/kg BID (Twice Daily Dosing); The analysis compares each of the 80 and 120 µg/kg BID groups with the untreated control group using analysis of covariance (ANCOVA), where the covariates are the baseline height SD score stratum used in the randomization, the pretreatment height velocity, the baseline bone age, the baseline chronological age, and sex; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 1.79, 95% CI [1.19 to 2.39], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Untreated vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 2.58, 95% CI [1.99 to 3.16], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: 80 μg/kg BID (Twice Daily Dosing) vs 120 μg/kg BID (Twice Daily Dosing); The analysis compares the 80 and 120 µg/kg BID groups using analysis of covariance (ANCOVA), where the covariates are the baseline height SD score stratum used in the randomization, the pretreatment height velocity, the baseline bone age, the baseline chronological age, and sex; Test type: Superiority or Other; p = 0.0032, ANCOVA; LS mean difference = 0.79, 95% CI [0.27 to 1.31], Standard Error of Mean 0.26

2. Secondary Outcome: Change From Baseline in Height Standard Deviation (SD) Score at One Year - ITT Population
Description: Height to be measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. Reposition subject between each measurement. Please note that Standard Deviation (SD) Score is a term used in growth studies. The SD Score is calculated as the patient value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child.
Time Frame: Measured at baseline and at one year
Population: A modified intention-to-treat population that consists of all randomized subjects in the untreated control, 80 and 120 µg/kg BID groups with a baseline height measurement and at least one on-treatment height measurement. Subjects assigned to 40 μg/kg BID arm were excluded from the analysis due to the dose change to 120 μg/kg BID.
Measure: Mean (Standard Deviation); unit: SD/year
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 22 | 0 | 42 | 49
SD/year | 0.02 (0.24) |  | 0.38 (0.17) | 0.48 (0.32)
Statistical Analysis 1: Comparison: Untreated vs 80 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 0.37, 95% CI [0.24 to 0.50], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Untreated vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 0.47, 95% CI [0.34 to 0.60], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: 80 μg/kg BID (Twice Daily Dosing) vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0495, ANCOVA; LS mean difference = 0.11, 95% CI [0.00 to 0.22], Standard Error of Mean 0.05

3. Secondary Outcome: Changes in Bone Age From Baseline to One Year
Description: Plain X-rays of the left hand and wrist exposed for bone age appraisal. The films are sent to a central facility for standardized evaluation.
Time Frame: Measured at baseline and at one year
Population: All randomized subjects in the untreated control, 80 and 120 µg/kg BID groups with baseline measurement and Month 12 measurement. Subjects assigned to 40 μg/kg BID arm were excluded from the analysis due to the dose change to 120 μg/kg BID.
Measure: Mean (Standard Deviation); unit: Year
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 23 | 0 | 40 | 44
Year | 0.8 (0.3) |  | 1.1 (0.4) | 1.2 (0.5)

4. Secondary Outcome: Percent Changes From Baseline in Serum Concentrations of IGF-1 at One Year
Description: Blood sample was collected while subject is in a fasting state for measuring the level of IGF-1 in the growth factor panel.
Time Frame: Measured at baseline and at one year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 18 | 0 | 34 | 42
Percent change | 64 (120) |  | 227 (220) | 266 (215)

5. Secondary Outcome: Percent Changes From Baseline in Serum Concentrations of IGF-2 at One Year
Description: Blood sample was collected for measuring the level of IGF-2 in the growth factor panel.
Time Frame: Measured at baseline and at one year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 17 | 0 | 35 | 40
Percent change | 14 (28) |  | -38 (37) | -37 (32)

6. Secondary Outcome: Percent Changes From Baseline in Serum Concentrations of Insulin-like Growth Factor Binding Protein-2 (IGFBP-2) at One Year
Description: Blood sample was collected for measuring the level of insulin-like growth factor binding protein-2 (IGFBP-2) in the growth factor panel.
Time Frame: Measured at baseline and at one year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 15 | 0 | 32 | 34
Percent change | -16 (26) |  | 58 (84) | 61 (79)

7. Secondary Outcome: Percent Changes From Baseline in Serum Concentrations of Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) at One Year
Description: Blood sample was collected while subject is in a fasting state for measuring the level of IGFBP-3 in the growth factor panel.
Time Frame: Measured at baseline and at one year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 18 | 0 | 34 | 42
Percent change | 13 (33) |  | -19 (22) | -19 (28)

8. Secondary Outcome: IGF Generation Test: Change of Serum IGF-1 After 7 Days Exposure to Recombinant Human Growth Hormone (rhGH)
Description: Blood drawn at Study Day 1, followed by 7 days of rhGH daily dosing at 0.05 mg/kg of body weight. Additional blood draw at Study Day 7.
Time Frame: Study Day 1 and Day 7
Population: All randomized subjects in the untreated control, 80 and 120 µg/kg BID groups with measurements both pre and post exposure to rhGH. Subjects assigned to 40 μg/kg BID arm were excluded from the analysis due to the dose change to 120 μg/kg BID.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 18 | 0 | 34 | 42
ng/mL | 40 (49) |  | 53 (49) | 48 (43)

9. Secondary Outcome: IGF Generation Test: Change of Serum IGFBP-3 After 7 Days Exposure to Recombinant Human Growth Hormone (rhGH)
Description: as for outcome 8
Time Frame: Study Day 1 and Day 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 18 | 0 | 34 | 42
mg/dL | 744 (459) |  | 800 (1095) | 681 (568)

10. Post Hoc Outcome: Height Velocity During the First Year for Subjects - Completers
Description: as for outcome 1
Time Frame: One Year
Population: All randomized subjects who completed 12 months of treatment in the untreated control, 80 and 120 µg/kg BID groups with a baseline height measurement and at least one on-treatment height measurement. Subjects assigned to 40 μg/kg BID arm were excluded from the analysis due to the dose change to 120 μg/kg BID.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 21 | 0 | 39 | 43
cm/year | 5.2 (1.0) |  | 7.0 (1.0) | 7.9 (1.4)
Statistical Analysis 1: Comparison: Untreated vs 80 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 1.83, 95% CI [1.26 to 2.40], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Untreated vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 2.83, 95% CI [2.26 to 3.39], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: 80 μg/kg BID (Twice Daily Dosing) vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0002, ANCOVA; LS mean difference = 1.01, 95% CI [0.50 to 1.51], Standard Error of Mean 0.25

11. Post Hoc Outcome: Change From Baseline in Height Standard Deviation (SD) Score at One Year - Completers
Description: as for outcome 2
Time Frame: One Year
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: SD/year
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Number analyzed (Participants) | 21 | 0 | 39 | 43
SD/year | 0.02 (0.24) |  | 0.39 (0.17) | 0.53 (0.30)
Statistical Analysis 1: Comparison: Untreated vs 80 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 0.37, 95% CI [0.25 to 0.50], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Untreated vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The two-sided p-values for the comparisons are adjusted for multiple comparisons using Dunnett's method; LS mean difference = 0.52, 95% CI [0.39 to 0.64], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: 80 μg/kg BID (Twice Daily Dosing) vs 120 μg/kg BID (Twice Daily Dosing); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0071, ANCOVA; LS mean difference = 0.15, 95% CI [0.04 to 0.26], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: Adverse events were collected until 30 days after last subject visit or until resolution. Adverse event collection for an individual subject was 1 year 1 month. Across study adverse event reporting continued for a total of 4 years 5 months.
Arm/Group | Untreated | 40 μg/kg BID (Twice Daily Dosing) | 80 μg/kg BID (Twice Daily Dosing) | 120 μg/kg BID (Twice Daily Dosing)
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/16 | 2/44 | 5/51
Other Adverse Events (participants affected / at risk) | 18/25 | 16/16 | 37/44 | 43/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Untreated (N=25) | 40 μg/kg BID (Twice Daily Dosing) (N=16) | 80 μg/kg BID (Twice Daily Dosing) (N=44) | 120 μg/kg BID (Twice Daily Dosing) (N=51)
Cor Triatriatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemic seizure (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis escherichia coli (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign Itracranial Hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Untreated (N=25) | 40 μg/kg BID (Twice Daily Dosing) (N=16) | 80 μg/kg BID (Twice Daily Dosing) (N=44) | 120 μg/kg BID (Twice Daily Dosing) (N=51)
Headache (Nervous system disorders) | 4 (9) | 8 (16) | 13 (30) | 21 (35)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 3 (5) | 10 (17) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (6) | 10 (17) | 7 (7)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (3) | 5 (5) | 7 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 3 (3) | 9 (10) — In order to avoid under-reporting hypoglycemia, transient symptoms with no accompanying blood glucose measurements were also reported as "hypoglycemia" or "hypoglycemia/decreased blood glucose".
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (4) | 8 (10) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 1 (1) | 4 (6) | 7 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 5 (6) | 5 (7)
Injection site bruising (General disorders) | 0 (0) | 3 (3) | 6 (10) | 4 (7)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 7 (7) | 4 (6)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 4 (7) | 7 (10)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 6 (7) | 2 (2)
Otitis media (Infections and infestations) | 3 (3) | 3 (3) | 2 (3) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (5) | 6 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4) | 4 (4)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 3 (4) | 4 (7) | 3 (4)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 1 (1) | 6 (8)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 4 (8)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator may publish or report data from their own subjects. The trial data in aggregate are the property of Tercica, Inc. and may not be published without permission of Tercica, Inc. Tercica, Inc. will be the final arbitrator of issues relating to the publication or presentation of the aggregate data.